CLINICAL TRIAL: NCT00656058
Title: Multi-Institutional Prospective Phase II Study of Montelukast for the Treatment of Bronchiolitis Obliterans Following Allogeneic or Autologous Stem Cell Transplantation in Children and Adults
Brief Title: Montelukast to Treat Bronchiolitis Obliterans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald Gress, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080097; 08-C-0097
Record Dates: First submitted 2008-04-09; First posted 2008-04-10 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Bronchiolitis Obliterans; Chronic Graft Versus Host Disease; Leukotriene; Montelukast; Stem Cell Transplant
Keywords: Leukotriene; Chronic Graft-Versus-Host Disease; Montelukast; Stem Cell Transplant; Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans; Bronchiolitis Obliterans Syndrome | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Montelukast to Treat Bronchiolitis Obliterans (Experimental): Montelukast for the treatment of BO following allogeneic or autologous stem cell transplant.
  Interventions: Drug: Singulair (Montelukast Sodium)

INTERVENTIONS:
Drug: Singulair (Montelukast Sodium) — Singulair (Montelukast Sodium):5-10 mg (weight based dosing) by mouth (PO) hour of sleep (HS)

SUMMARY:
Background:

Bronchiolitis obliterans is a form of chronic graft-versus-host disease (GVHD) that sometimes develops after stem cell transplantation (SCT) or bone marrow transplantation (BMT).

In bronchiolitis obliterans, immune cells that normally fight infections attack the lungs of the transplant recipient, causing destruction of lung tissue and fibrosis (scarring). When fibrosis develops, the lungs cannot work properly.

Montelukast (Singulair) is a drug that has been used for many years to treat asthma. Its use as a treatment for bronchiolitis obliterans is experimental.

Objectives:

To see if montelukast improves or stabilizes lung function in patients who develop bronchiolitis obliterans after BMT or SCT.

To assess the safety of montelukast in patients with bronchiolitis obliterans after BMT or SCT

To see if montelukast affects the cells that damage the lungs.

To see if montelukast improves other forms of chronic GVHD, quality of life, and overall survival in patients with bronchiolitis obliterans after BMT or SCT.

Eligibility:

Patients 6 years of age and older with bronchiolitis obliterans following stem cell transplantation.

Design:

Patients take one montelukast tablet daily for 6 months and undergo the following procedures during this period:

* Lung function tests. The patient breathes into a machine that measures the amount of air that goes into and out of the lungs. This test is done once a month for 3 months, then at 6 months, 12 months and 24 months.
* Medical history and physical examination at the study site about every 3 months for the first year of the study and then at 12 months and 24 months. Patients also have physical examinations monthly for the first 6 months at their primary doctors office. Tests may include blood and urine tests, chest computed tomography (CT) scans, echocardiogram (heart ultrasound), 2- and 6-minute walk tests, and quality-of-life questionnaires.
* Bronchoalveolar lavage in patients 18 years of age and older. The subject s mouth, nose and airways are numbed with lidocaine. Some patients may need sedation or anesthesia for the procedure. A tube (bronchoscope) is then passed through the nose into the airway, and a small amount of fluid is put into the lung. The fluid is then removed and tested for infections or other lung problems.
* Apheresis to collect white blood cells. Whole blood is collected through a tube inserted into a vein in the arm. The white cells are extracted in a cell separator machine, and the rest of the blood is returned to the body through a tube placed in a vein in the other arm. The cells are used to study GVHD and bronchiolitis obliterans.
* Patients who wish to continue montelukast therapy after 6 months may do so under the care of their primary doctor, if both agree to the continuation....

DETAILED DESCRIPTION:
Background:

Bronchiolitis obliterans (BO) is an insidious disease with high mortality following allogeneic blood or marrow transplantation (BMT). There are no consistently effective treatments for BO following BMT and the pathogenesis is largely unknown.

The mechanisms underlying similar immune-mediated lung destructive processes are better elucidated. Rejection following allogeneic lung transplantation and scleroderma lung disease result from analogous immunologically mediated destruction of lung tissue leading to similar pathologic and clinical presentations to post-BMT BO.

Increased leukotriene production has recently been implicated in the development of both post-lung transplant BO and scleroderma lung disease in animal models and patient studies.

Montelukast (singulair) is an approved, well-tolerated, oral agent that inhibits leukotriene action in lung inflammation. This agent has been extensively used in children and adults to treat asthma with an excellent safety profile.

Objectives:

To evaluate if montelukast stabilizes or improves pulmonary function in patients with BO after BMT using forced expiratory volume 1 (FEV-1) changes as primary endpoints, and oxygen saturation, pulmonary function test (PFT) parameters (forced expiratory flow (FEF) 25-75, residual volume (RV) and RV/forced vital capacity (FVC), carbon monoxide diffusing capacity (DLC02), FEV-1/FVC, FEV-1/slow vital capacity (SVC) ratio), and timed walk tests as secondary endpoints.

To evaluate the safety of montelukast in the population of patients with BO after BMT.

To investigate if leukotriene elevation contributes to the pathogenesis of BO after BMT by measuring leukotriene levels of the blood, urine, and bronchoalveolar lavage (BAL), and leukotriene surface receptor expression on immune cells before and after montelukast administration.

To determine if montelukast improves other chronic graft versus host disease (cGVHD) manifestations, quality of life, and overall survival.

Eligibility:

Patients greater than or equal to 6 years old with bronchiolitis obliterans following stem cell transplantation for any disease indication may be enrolled.

Design:

This is a prospective phase II study, the primary aim of which is to assess whether montelukast improves or stabilizes the pulmonary function of patients with BO after BMT.

Primary outcome data will be analyzed in 2 ways. 1) The proportion of patients with stable or improved percent predicted of FEV-1 will be compared against benchmark data obtained from a literature review. 2) The slope of FEV-1 before and after the introduction of montelukast will be compared.

Pediatric and adult patients with BO following BMT will receive approved doses of montelukast continuously.

The planned length of the study would be 2 years per patient with primary endpoint at 6 months, permitting sufficient time to determine safety and meet other endpoints.

This phase II trial will be conducted at 2 institutions: National Institutes of Health (NIH) and Fred Hutchinson Cancer Research Center. Forty-five patients will be enrolled on this trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than 6 years old.

Diagnosis of bronchiolitis obliterans after allogeneic or autologous stem cell transplant. The criteria will be based on the definitions created by the National Institutes of Health (NIH) consortium on chronic graft versus host disease (cGVHD). As part of these criterion, for patients without pathologic evidence of BO, one other sign of chronic GVHD must be present. For diagnosis of cGVHD, a minimum of the following must be present: 1) a process distinct from that diagnosed as acute GVHD, 2) the presence of a diagnostic sign or a distinctive sign supported by another clinical or laboratory test, and 3) the exclusion of other pathologies (i.e. recurrent cancer, drug reaction or infection (see Appendix 5a for a list of diagnostic signs.). To meet criteria for a diagnosis of bronchiolitis obliterans, patients must fulfill all 3 criteria. Prior lung tissue biopsy will be analyzed and confirmed to show evidence of bronchiolitis obliterans by the National Cancer Institute (NCI) Laboratory of Pathology if available. If tissue is not available for confirmation, a new biopsy will not be performed.

For bronchiolitis obliterans:

1. Forced expiratory volume 1 (FEV1) less than or equal to 75 percent of predicted by pulmonary function evaluation for height and weight.
2. Evidence of air-trapping or small airway thickening or bronchiectasis on high resolution chest computed tomography (CT) and residual volume (RV) or RV/forced vital capacity (FVC) greater than 120 percent and evidence of chronic GVHD of another organ, OR FEV1/ vital capacity (slow or forced VC whichever is larger) ratio less than 5 percent of predicted for age or less than 0.7, OR pathologic evidence of bronchiolar inflammation and obstruction of the lumen consistent with a diagnosis of BO. Pulmonary function tests will utilize body plethysmography not helium studies for pertinent values when there is a discrepancy if available.
3. Absence of active infection with appropriate investigation of any clinical symptoms to include radiographic, microbiologic, and pathologic studies as determined by the PI or LAI.

   Patients must also have 2 PFT measurements with documented FEV1 values greater than 3 months apart to calculate the entry FEV1 slope. All available prior PFTs will be utilized for baseline slope calculation. For adult patients, the absolute FEV1 will be utilized for slope calculation; for pediatric patients, the percent predicted will be used. For patients enrolled after an acute decline following BMT without 2 post-BMT values greater than 3 months apart, the pre-BMT value may be utilized as the first value and the entry PFT value may be the second for the slope calculation. The baseline and 6th-cycle PFT should be done at the accruing site.

   Prior therapy: For patients with a chronic diagnosis of BO who have been on treatments, any prior therapy that has been administered chronically for > 3 months will be acceptable for enrollment as long as the patient has not demonstrated consistent improvement attributed to these agents in a one month (or more) period of observation preceding enrollment. For patients on steroids, a steroid burst exceeding and increase of one half mg/kg/day will be considered for the start of the 3 month monitoring period. Notably, documented intercurrent infections that are treated with antimicrobials that result in improvements to, but not above previous baselines will not be considered an improvement attributable to immunosuppressive therapy. Patients who have had consistent improvements in the months preceding trial entry will not be eligible since there will be no way to discern improvement due to montelukast versus another therapy. Alternatively, a patient with a new diagnosis of bronchiolitis obliterans characterized by a new decrease in FEV1 is also eligible for this study. Notably, patients who have received bronchodilators or other pulmonary therapies may be included in this study as long as montelukast is not part of this regimen.

   Performance status: Karnofsky or Lansky performance status greater than or equal to 40 percent (Appendix 1).

   Ability to give informed consent. For patients less than 18 years of age, their legal guardian must give informed consent. Pediatric patients will be included in an age appropriate discussion in accordance with NIH guidelines or participating institutional guidelines.

   Hepatic function: Patients must have evidence of adequate liver function prior to enrollment defined by total bilirubin less than 3 times the upper limit of normal and transaminases less than 5 times the upper limit of normal for age appropriate indices.

   Cardiac function: Patients must have evidence of adequate cardiac function prior to enrollment defined by ejection fraction greater than 25 percent performed within the last 6 months at NIH and absence of symptoms of cardiac disease at FHCRC, JHH, or Hackensack.

   Pulmonary function: Patients must have an FEV1 greater than or equal to 20 percent predicted for inclusion in this study.

   EXCLUSION CRITERIA:

   Underlying disease status: Patients with tumor burden greater than minimal residual disease (i.e. tumor burden that can only be detected by molecular methods) would be excluded from this study.

   Prior post-transplant treatment with montelukast or zakirlukast within the past 2 months and total duration of therapy does not exceed 3 months.

   Clinically significant systemic illness with manifestations of significant organ dysfunction which in the judgment of Principal or Associate Investigator would render the patient unlikely to tolerate the protocol therapy or complete the study.

   Patients must have been on their current cGVHD therapeutic regimen for at least 3 months with stable or decreasing FEV1 to be eligible for this trial. Any patient who has been on a therapy for less than 3 months for cGVHD will need to be monitored for 3 months without improvement in FEV1 prior to enrollment.

   Ventilated patients are excluded.

   Patients taking rifampin or phenobarbital as these medications alter the metabolism of montelukast.

   Patients taking greater than one age-appropriate dose of ibuprofen or aspirin containing products per day that inhibit cyclooxygenase will be excluded from this trial. The acceptable upper limit for adult daily doses of aspirin is 650mg/day and 800mg/day of ibuprophen. For children, the acceptable upper limit of ibuprophen is pediatric dose per day (less than 10 mg per kg to a maximum of 800 mg). Children should not take aspirin due to risk of Reye's syndrome unless specifically prescribed by their physician.

   Patients with a history of allergy to montelukast.

   Pregnant females and nursing mothers will be excluded from this trial due to unknown risks to the developing fetus. While on study, patients of child-bearing potential must be able to consent to utilize effective birth control measures.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06-17 (Actual); Primary Completion 2014-05-02 (Actual); Study Completion 2018-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Gress, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams KM, Hnatiuk O, Mitchell SA, Baird K, Gadalla SM, Steinberg SM, Shelhamer J, Carpenter A, Avila D, Taylor T, Grkovic L, Pulanic D, Comis LE, Blacklock-Schuver B, Gress RE, Pavletic SZ. NHANES III equations enhance early detection and mortality prediction of bronchiolitis obliterans syndrome after hematopoietic SCT. Bone Marrow Transplant. 2014 Apr;49(4):561-6. doi: 10.1038/bmt.2013.222. Epub 2014 Jan 13. PMID 24419526
- [Result] Oral presentation: "Interim Analysis of a Phase II Trial of Montelukast for the Treatment of Bronchiolitis Obliterans Syndrome after HSCT reveal Immunobiology of Disease American Society of Blood and Marrow Transplantation 2013
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0097.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Montelukast to Treat Bronchiolitis Obliterans: Montelukast for the treatment of BO following allogeneic or autologous stem cell transplant.
  Singular (Montelukast Sodium): Singular (Montelukast Sodium):5-10 mg (weight based dosing) PO HS
Period: Overall Study
Arm/Group | Montelukast to Treat Bronchiolitis Obliterans
Started | 25
Completed | 19
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Montelukast to Treat Bronchiolitis Obliterans
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 23
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.29 (15.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stable or Improved Predicted Forced Expiratory Volume 1 (FEV-1) With Published Literature
Description: Responsive disease (RD) will be defined as ≥15% absolute improvement in the percentage predicted FEV-1. Progressive disease (PD) will be defined as >15% decrease in FEV-1 documented on 2 pulmonary function test (PFT) evaluations greater than 2 weeks apart. Stable disease (SD) will be defined as <15% change in the absolute FEV-1.
Time Frame: 180 days
Population: No data is available for the one missing participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast to Treat Bronchiolitis Obliterans
Number analyzed (Participants) | 19
Participants
  Increased 5-13% of predicted | 5
  Stable | 7
  Declined | 6
  Missing | 1

2. Primary Outcome: Number of Participants With Improved, Stable or Declined Forced Expiratory Volume 1 (FEV-1) Slope at 6 Months
Description: FEV-1 slope of decline was generated using regression line of FEV-1 value vs. days post hematopoietic stem cell transplant. Responsive disease (RD) for the slope of FEV-1 change will be an increase in the slope of absolute FEV-1. Progressive disease (PD) for the slope of FEV-1 change will be a decrease in the slope of absolute FEV-1. Stable disease (SD) for the slope of FEV-1 change will be a 0 change in FEV-1 slope.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast to Treat Bronchiolitis Obliterans
Number analyzed (Participants) | 19
Participants
  Improved | 9
  Stable | 9
  Declined | 1

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 71 months and 17 days
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast to Treat Bronchiolitis Obliterans
Number analyzed (Participants) | 25
Participants | 20

4. Secondary Outcome: Forced Expiratory Volume 1 (FEV-1)/Vital Capacity (VC)
Description: Pulmonary function test performed for eligibility and baseline.
Time Frame: Baseline
Measure: Median (Full Range); unit: Ratio
Arm/Group | Montelukast to Treat Bronchiolitis Obliterans
Number analyzed (Participants) | 19
Ratio | 0.5 [0.29 to 0.78]

5. Secondary Outcome: Percentage Overall 2-Year Survival
Description: Percentage of participants alive at 2 years.
Time Frame: 2 years
Population: This is a multicenter study and the number analyzed reflect data for evaluable subjects enrolled at the National Institutes of Health only.
Measure: Number; unit: percentage of participants
Arm/Group | Montelukast to Treat Bronchiolitis Obliterans
Number analyzed (Participants) | 12
percentage of participants | 84

6. Secondary Outcome: Number of Non-Infected Participants at Baseline With Cysteinyl Leukotriene Receptor Expression on Cluster of Differentiation (CD4) and CD8 T Cells, Granulocytes, and Eosinophils in Bronchoalveolar Lavage (BAL) Fluid
Description: Fluid from the bronchoalveolar lavage in adult participants (pediatric optional) will be collected and sent to the lab to be evaluated for infectious diseases by flow cytometry
Time Frame: Day 1 of study
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast to Treat Bronchiolitis Obliterans
Number analyzed (Participants) | 19
Participants | 19

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 71 months and 17 days.
Description: The serious adverse events while on study are not possibly, probably, or definitely related to montelukast or attributed to research interventions.
Arm/Group | Montelukast to Treat Bronchiolitis Obliterans
All-Cause Mortality (participants affected / at risk) | 3/25
Serious Adverse Events (participants affected / at risk) | 15/25
Other Adverse Events (participants affected / at risk) | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast to Treat Bronchiolitis Obliterans (N=25)
Anorexia (Gastrointestinal disorders) | 1 (1)
Death not associated with CTCAE term::Death NOS (General disorders) | 2 (2)
Death not associated with CTCAE term::Multi-organ failure (General disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Gastrointestinal - Other (gastroenteritis) (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI::Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infection - Other (CMV reactivation) (Infections and infestations) | 1 (2)
Infection - Other (pneumonia/infection with unknown ANC) (Infections and infestations) | 1 (1)
Infection - Other (sinusitis) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 4 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 1 (4)
Infection with unknown ANC::Colon (Infections and infestations) | 1 (1)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 1 (1)
Joint-effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Mood alteration::Depression (Nervous system disorders) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Parainfluenza Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RSV Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast to Treat Bronchiolitis Obliterans (N=25)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (5)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 4 (5)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (5)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1)
Gastrointestinal - Other (Pneumatosis coli) (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Hemorrhage, pulmonary/upper respiratory::Lung (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection - Other (Helicobacter pylori infection) (Infections and infestations) | 1 (1)
Infection - Other (S. Maltophilia) (Infections and infestations) | 1 (1)
Infection - Other (URI) (Infections and infestations) | 1 (1)
Infection - Other (Viral infection (evaluated by home physicians)) (Infections and infestations) | 1 (1)
Infection - Other (fever and URI symptoms) (Infections and infestations) | 1 (2)
Infection - Other (upper respiratory infection) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 2 (2)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with unknown ANC::Sinus (Infections and infestations) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Lipase (Metabolism and nutrition disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Nervous system disorders) | 1 (1)
Pain::Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4 (5)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (URI) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Renal/Genitourinary - Other (interstitial renal fibrosis) (Renal and urinary disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Weight loss (General disorders) | 2 (2)
Pain: joint (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT00656058/Prot_ICF_000.pdf